CLINICAL TRIAL: NCT06981351
Title: Matching Treatments to Cognitive Deficits in Offenders With Substance Use Disorders
Acronym: MCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Mind Research Network (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24615; R01DA058004 (NIH)
Record Dates: First submitted 2025-04-24; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: Antisocial Behavior
Keywords: Cognitive skills training; Attention to Context; Affective Cognitive Control
MeSH Terms: conditions — Antisocial Personality Disorder

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Staff that conduct cognitive skills training sessions will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Attention to context deficit (Experimental): Participants with attention to context deficits will receive treatment either targeted towards their specific deficit (matched) or towards affective cognitive control deficits (mismatched).
  Interventions: Behavioral: Attention to Context (ATC) training; Behavioral: Affective Cognitive Control (ACC) training
- Affective Cognitive Control deficit (Experimental): Participants with affective cognitive control deficits will receive treatment either targeted towards their specific deficit (matched) or towards attention to context deficits (mismatched).
  Interventions: Behavioral: Attention to Context (ATC) training; Behavioral: Affective Cognitive Control (ACC) training
- No psychopathology (Experimental): Participants in the no psychopathology group will receive one of the two treatment types (ATC or ACC).
  Interventions: Behavioral: Attention to Context (ATC) training; Behavioral: Affective Cognitive Control (ACC) training

INTERVENTIONS:
Behavioral: Attention to Context (ATC) training — ATC training focuses on learning to attend to and integrate contextual cues present in the environment. Three tasks, Reversal Learning, Divided Visual Field, and Affective Gaze, require ATC functioning and provide individuals with practice noticing changes in contextual information, such as rule changes and using emotion information to modulate behavior.
Behavioral: Affective Cognitive Control (ACC) training — ACC training focuses on providing individuals with practice inhibiting behavior, particularly within motivational or affective contexts. Three tasks, Shapes, Numbers, and Lottery, tap ACC functioning and place demands on the basic employment of cognitive control, such as task switching, as well as on the concurrent engagement of cognitive control and affective processing.

SUMMARY:
The goal of this clinical trial is to investigate the effect of two types of cognitive remediation training on real-world behavioral outcomes including substance use, institutional adjustment, and recidivism following release from prison. Each training type is designed to target one of two subtypes of antisocial criminal offenders, who are characterized by either: 1) Attention to context-based deficits, or 2) Affective cognitive control-based deficits.

The main questions it aims to answer are:

Does matching deficit type with targeted cognitive training improve outcomes (relative to mismatched training)? What are the functional brain mechanisms that underlie treatment change?

Participants will:

Be assigned to cognitive training that either does or does not match their deficit type.

Complete six one-hour sessions of cognitive skills training. Complete pre and post-training behavioral tasks assessing self-regulation deficits.

Complete structural MRI scans and functional MRI scans assessing cognitive control.

Complete post-treatment follow-up assessments evaluating self-regulation, adjustment, and stressful life events, substance use and recidivism.

DETAILED DESCRIPTION:
Prior research has identified two subtypes of antisocial offenders, typified by distinct dysfunctional cognitive emotion interactions undermining self-regulation. One subtype is characterized by an attention-based abnormality, which impairs adaptive processing of contextual information, tangential to one's primary focus. This abnormality is typified by offenders with high levels of callous/unemotional traits. A second subtype is characterized by hyper-reactions to personally relevant cues, interfering with executive functions that are otherwise needed to regulate behavior. This abnormality is prevalent in those with high externalizing characteristics. The investigators have developed cognitive skills training that addresses each of these specific deficits in distinct ways. These distinct interventions are intended to address mechanism-specific cognitive emotional dysfunction, as opposed to treating distinct dysfunctions with a uniform approach. The investigators' NIH-funded pilot work has shown evidence of improving outcomes in offenders by matching specific deficits with focused skills training. This project will execute a well-powered, randomized clinical trial to demonstrate reliability and generalizability of these effects. We expect to verify prior findings of improved outcomes by matching individual deficits with the targeted interventions. Effects of treatment on specific cognitive skills (assessed by laboratory-based tests) and real-world behavioral outcomes including substance use behaviors, institutional adjustment, and recidivism following release from prison will be examined. Further, advanced neuroimaging measures will be used to assess brain changes with treatment. This will aid in specifying potentially different mechanisms of treatment success in each respective group. This project addresses the ongoing need to improve and validate focused interventions that target specific deficits, replacing less-effective one-size-fits-all approaches.

ELIGIBILITY:
Inclusion Criteria:

* Currently incarcerated
* No uncorrectable auditory or visual deficits
* Able to speak and/or understand English
* 5th grade reading level or higher
* IQ score = 80 or above
* Lifetime history of substance use disorder based on DSM criteria
* No history of dementia or other cognitive disability
* No indication of current psychotic disorder
* No major medical illness or CNS disease
* Scores from the Psychopathy Checklist-Revised (PCL-R) meet criteria for one of the designated treatment groups

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Biological sex at birth is male
Enrollment: 288 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive task performance - Stroop | From enrollment to end of treatment at six weeks
  Stroop task. Performance is quantified by number of correct responses (0 - 100)%.
Cognitive task performance - Lexical Decision Making | From enrollment to end of treatment at six weeks
  Lexical Decision Making task. Performance is quantified by number of correct responses (0 - 100%).
Cognitive task performance - Delay Discounting | From enrollment to end of treatment at six weeks
  Delay Discounting task. Performance is quantified quantified by calculating where the answers place the respondent amid reference discounting curves. Range 0.0-0.5.
Functional MRI - Go/NoGo task performance | Change assessed from enrollment to end of treatment at six weeks
  Functional MRI task performance (Go/NoGo task). Performance is quantified by the number of 'false alarms' (responding to the NoGo stimulus). Range 0-39.
Functional MRI - Go/Nogo brain response | Activity assessed during MRI scan. Change assessed from enrollment to end of treatment at six weeks
  Change (i.e. increased or decreased) in functional brain response (Blood Oxygen Level Dependent/BOLD) in region of interest (anterior cingulate) assessed using Statistical Parametric Mapping (SPM).
Real-World Outcomes - Substance use (TLFB) | From enrollment to six months post-release from incarceration
  Substance use. Assessed using the timeline follow back (TLFB) - calendar recording dates of use for stimulant drugs.
Real-World Outcomes - Substance use (ASE) | From enrollment to six months post-release from incarceration
  Substance use. Assessed using the Abstinence Self Efficacy scale (higher scores indicate greater difficulty with abstinence). Range 0-4.
Real-World Outcomes - Substance use (DUDIT) | From enrollment to six months post-release from incarceration
  Substance use. Assessed using the Drug Use Disorders Identification test (higher scores indicate more/severe substance use). Range 0-44.
Real-World Outcomes - Criminal behavior | From enrollment to six months post-release from incarceration
  Criminal behavior. Assessed using the Crime Inventory - records the number of instances of criminal behavior
Risky Impulsive Self-Destructive Behavior | From enrollment to six months post-release from incarceration
  The RISQ questionnaire measures risky, impulsive, and self-destructive behaviors in 8 domains (aggression, self-harm, gambling, impulsive spending/driving, impulsive eating, risky sex, illegal behavior, and alcohol use). For each behavior, respondents note the number of times they have engaged in the behavior in their lifetime. Higher scores indicate more severe risky, impulsive, and self destructive behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Mind Research Network/Lovelace Biomedical Research Institute, Albuquerque, New Mexico, United States